CLINICAL TRIAL: NCT01384110
Title: Efficacy of a Brown Seaweed Extract Rich in Polyphenols on Glycemic Response to Sucrose in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: innoVactiv Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2010-RD-01-CLN
Record Dates: First submitted 2011-06-13; First posted 2011-06-28 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Hyperglycemia
Keywords: Amylase; Glucosidase; Glycemic response; Sucrose; Seaweed
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brown Seaweed Lemon Tea (Experimental): Single administration of lemon tea containing 500 mg of brown seaweed powder and 50 g of sucrose
  Interventions: Dietary Supplement: Reduction of glycemic index of ingested foods
- Placebo lemon tea (Placebo Comparator): Single administration of placebo lemon tea containing 50 g of sucrose
  Interventions: Dietary Supplement: Reduction of glycemic index of ingested foods

INTERVENTIONS:
Dietary Supplement: Reduction of glycemic index of ingested foods — Oral administration of the experimental lemon tea powder(56.1 g) and the placebo lemon tea powder (55.6 g) dissolved in water. Each participant will receive both treatment in a cross-over protocol design during 2 visits separated by a 2-weeks period. The day before both intervention, participants will consume a standardised meal for the supper.
  Other Names: InSea2

SUMMARY:
The primary endpoint of this trial will be to evaluate if a single administration in human of a lemon ice tea containing 500 mg of a polyphenol-rich algal powder is able to reduce postprandial glycemia and insulinemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 18 to 60
* BMI between 20 and 30
* Non-smoking
* Using valid contraceptive method (women of childbearing age)

Exclusion Criteria:

* Iodine allergy, or allergy to components of the test product or placebo or standard meal
* Diabetes
* Use of dietary supplements for duration of study
* History of gastro-intestinal affections, anemia, major surgeries or surgeries of the stomach or digestive tract

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Significant reduction in postprandial glycemia | Immediately after product administration (single use)
Significant reduction in postprandial insulinemia | Immediately after product administration (single use)

SECONDARY OUTCOMES:
Frequency and severity of Adverse Events as a Measure of Safety and Tolerability | First administration up to 7 days after last administration

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, Principal Investigator — Institut des nutraceutiques et des aliments fonctionnels
Locations (1):
- Institut des Nutraceutiques et des Aliments Fonctionnels (INAF), Québec, Quebec, Canada